CLINICAL TRIAL: NCT04961034
Title: Peri Kasai Portoenterostomy Anchoring of the Jejunal Loop
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mohammad Gharieb Mohammad Khirallah, Associate professor of pediatric surgery, Tanta University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 33943/7/20
Record Dates: First submitted 2021-07-09; First posted 2021-07-14 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Biliary Atresia
Keywords: biliary atresia; kasai portoenterostomy; modified; cholangitis
MeSH Terms: conditions — Biliary Atresia; Cholangitis | interventions — Portoenterostomy, Hepatic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- classic KPE (Other): the classic management of biliary atresia as described
  Interventions: Procedure: kasai portoenterostomy
- modified KPE (Other): we added 2 sutures posterior, one on each side and two anterior. this will hang the jejunal loop to promote tension free anastomosis
  Interventions: Procedure: kasai portoenterostomy

INTERVENTIONS:
Procedure: kasai portoenterostomy — surgical creation of stoma between porta hepatis and jejunal loop

SUMMARY:
the study of the effect o the hanging of the jejunal loop to the peri KPE Glisson capsule on the rate of bile drainage and requirement of liver transplantation

DETAILED DESCRIPTION:
To evaluate the effect of anchoring jejunal loop to Glisson capsule of liver after completion of modified Kasai portoenterostomy (KPE) on the frequency of attacks of cholangitis and the overall incidence of native liver survival.

Methods: Retrospective study included 29 infants diagnosed as biliary atresia (BA). They were subjected to modified KPE. Two subgroups were present. Group A included 16 infants and had KPE. Group B included 13 infants and had the assumed modification. Wider dissection of fibrous portal plate was considered in both groups. After completion of KPE, the jejunal loop anchored to Glisson capsule of liver at porta hepatis in group B.

ELIGIBILITY:
Inclusion Criteria:

* infants with biliary atresia diagnosed and treated before 60th day of age

Exclusion Criteria:

* infants older than 60 days

Ages: 4 Weeks to 8 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 26 (Estimated)
Dates: Start 2015-01 (Actual); Primary Completion 2021-06 (Actual); Study Completion 2023-12-20 (Estimated)

PRIMARY OUTCOMES:
the total number of cholangitis | two years
  the total attacks of chollangitis
number of native liver survivors | two years
  the decrease of the need of liver transplantation in children with biliary atresia

SECONDARY OUTCOMES:
early improvement of liver functions | 6 months
  normalization of liver function

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Tanta University, Tanta, Gharbia Governorate
  - Tantra Universiy, Tanta

IPD SHARING:
Plan to Share IPD: Yes
publication as article
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 6 months